CLINICAL TRIAL: NCT03352180
Title: Do Concomitant Subscapularis Tears in Large to Massive Rotator Cuff Tears
Brief Title: Subscapularis Tears in Large to Massive Rotator Cuff Tear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Woo Kim, Department of Orthopedic Surgery, Wonkwang University Hospital, Iksan, Korea Professor Jeong Woo Kim, MD, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201608-HR091
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Massive Rotator Cuff Tears

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- subscapularis tendon repair (Active Comparator): arthroscopic reapir of subscapularis tendon
  Interventions: Procedure: arthroscopic reapir of subscapularis tendon
- subscapularis tendon debridement (Active Comparator): arthroscopic debredement of subscapularis tendon
  Interventions: Procedure: arthroscopic debridement of subscapularis tendon

INTERVENTIONS:
Procedure: arthroscopic reapir of subscapularis tendon — arthroscopic reapir of massive rotator cuff tears involving the subscapularis.
  Arms: subscapularis tendon repair
Procedure: arthroscopic debridement of subscapularis tendon — arthroscopic debridement of massive rotator cuff tears involving the subscapularis.
  Arms: subscapularis tendon debridement

SUMMARY:
Do concomitant subscapularis tears in large to massive rotator cuff tears affect postoperative functional and structural outcomes?

Background and purpose:

The subscarpularis tendon is essential force maintaining normal glenohumeral biomechanics. However, there are few studies which have addressed the outcomes of tears extending to the subscapularis tendon in massive rotator cuff tears. The purpose of this study was to assess the clinical and structural outcomes of arthroscopic reapair of massive rotator cuff tears involving the subscapulrais.

DETAILED DESCRIPTION:
MATRALS AND METHODS This retrospective comparative study was approved by our institutional review board.

Patient Selection This study targeted patients who had undergone arthroscopic rotator cuff repair, which was performed by a single surgeon in our institution between January 2010 and January 2014.

The inclusion criteria were as follows: (1) a full-thickness superoposterior rotator cuff tear larger than 5 cm(19) or complete superoposterior rotator cuff tear(24) identified on preoperative MRI and intra operative arthroscopic findings, (2) a follow-up MRI evaluation at 6 months after surgery, and (3) a clinical assessment performed a minimum 2 years postoperatively. The exclusion criteria were as follows: (1) small, medium, or large tears(21); (2) a partial-thickness tear; (3) an isolated subscapularis tear; (4) failure of subscapularis repair at the time of the index procedure; (5) previous rotator cuff surgery of the affected shoulder; (6) concomitant surgery for glenohumeral joint instability or other bony procedure; and (7) substantial glenohumeral arthritis (Hamada classification29 grade 4) or inflammatory arthropathy of the affected shoulder.

Tear Classification Rotator cuff tear patterns were classified into the following 3 categories according to the tear size of the subscapularis tendon on preoperative MRI: I-massive tear, intact subscapularis tendon; S-massive tear, tear involving half or less than half of the subscapularis tendon; and L-massive tear, tear extending to more than half of the subscapularis tendon.

Clinical Assessments Clinical data were recorded on the day before surgery and at final follow-up (at least 24 months postoperatively) by fellowship trainees. Four outcome measures were used in this study: VAS pain score, ASES score, Constant score, and active shoulder ROM. The ASES score involves a score summation using a 100-point system (50 points for daily function and 50 points for pain).

Radiographic Evaluation A standard set of plain radiographs was obtained as follows: anteroposterior (AP) views in internal rotation and external rotation, supraspinatus outlet view, axillary view, and Rockwood view (30 caudally angled AP view). We evaluated fatty degeneration of the rotator cuff muscle preoperatively with MRI, using the 5-stage grading system27: grade 0, no fatty deposit; grade 1, some fatty streaks; grade 2, more muscle than fat; grade 3, as much muscle as fat; and grade 4, less muscle than fat. The integrity of rotator cuff repair was determined by ultrasonographic evaluation. All patients underwent a postoperative ultrasonographic examination at 4.5 months and 12 months or later after surgery. One specialized radiologist with more than 10 years of experience in musculoskeletal ultrasonography performed all follow-up examinations using an HDI 5000 system or an IU-22 system (both from Philips Healthcare). He did not receive any information on intraoperative findings and subsequent operative procedures. An ultrasonographic evaluation of the rotator cuff was performed according to the standard protocol.42 The ultrasound criteria for the diagnosis of full-thickness rotator cuff tears were as follows5,54: (1) absence of observation of the supraspinatus tendon attributable to retraction under the acromioclavicular joint; (2) localized absence or focal discontinuity of the rotator cuff with concomitant loss of the normal anterior arc of the subdeltoid bursa; (3) loss of the normal supraspinatus substance with widening of the gap between the supraspinatus and biceps tendons, including exposure of a bare area of bone and cartilage; (4) a hypoechoic or anechoic cleft extending through the entire substance of the rotator cuff; and (5) coexistence of fluid in the subacromial-subdeltoid bursa and/or presence of fluid in the sheath of the long head of the biceps tendon. Partialthickness tears were diagnosed based on the presence of a focal hypoechoic or anechoic defect in the tendon, involving either the bursal or articular surface and manifesting in 2 perpendicular planes.54

ELIGIBILITY:
Inclusion Criteria:

1. a full-thickness superoposterior rotator cuff tear larger than 5 cm or complete superoposterior rotator cuff tear identified on preoperative MRI and intra operative arthroscopic findings
2. a follow-up MRI evaluation at 6 months after surgery, and
3. a clinical assessment performed a minimum 2 years postoperatively.

Exclusion Criteria:

1. small, medium, or large tears
2. a partial-thickness tear
3. an isolated subscapularis tear
4. failure of subscapularis repair at the time of the index procedure
5. previous rotator cuff surgery of the affected shoulder
6. concomitant surgery for glenohumeral joint instability or other bony procedure
7. substantial glenohumeral arthritis (Hamada classification grade 4) or inflammatory arthropathy of the affected shoulder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-07-11 (Estimated); Study Completion 2019-07-11 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 4weeks
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.

SECONDARY OUTCOMES:
The American Shoulder and Elbow Surgeons Shoulder Score (ASES) | 4weeks
  reliability, validity, and responsiveness

CONTACTS AND LOCATIONS:
Locations (1):
- Wonkwang University Hospital, Iksan, Jeollabuk-do, South Korea